CLINICAL TRIAL: NCT06428045
Title: Synergistic Treatment With Antiretrovirals and Laser Interstitial Thermal thErapy (STARLITE) for Unresectable High-Grade Gliomas: A Phase 1 Study
Brief Title: STARLITE for Unresectable High-Grade Gliomas
Acronym: STARLITE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ashish Shah, Assistant Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20231163
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: High Grade Glioma
Keywords: Unresectable High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy; abacavir; Lamivudine; Ritonavir; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation/de-escalation and dose expansion design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Part 1: STARLITE Dose Escalation/De-Escalation Cohort (Experimental): Participants in this group will undergo Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MR-guided LITT) on Day 0 after stereotactic needle biopsy. On Day 7, participants will begin combination antiretroviral therapy (ART) consisting of Abacavir, Lamivudine, and dose escalation/de-escalation of Ritonavir (RTV), to determine the recommended Phase 2 dose (RP2D) of Ritonavir. Participants will receive up to 12 months of ART.
  Beginning Day 14 through Day 180, participants will receive adjuvant therapy, standard of care consisting of focal radiotherapy and Temozolomide therapy. Participants will receive focal radiotherapy for six weeks (42 days). Participants will be administered Temozolomide up to Day 180.
  Participants will receive up to 12 months of study therapy, followed by up to 12 months of follow-up. Total participation duration is up to 24 months.
  Interventions: Procedure: Magnetic Resonance (MR)-guided Laser Interstitial Thermal Therapy (LITT); Drug: Abacavir; Drug: Lamivudine; Drug: Ritonavir; Drug: Temozolomide; Radiation: Focal Radiotherapy
- Part 2: STARLITE Dose Expansion Cohort (Experimental): Participants in this group will undergo Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MR-guided LITT) after biopsy on Day 0. On Day 7, participants will begin combination antiretroviral therapy (ART) consisting of Abacavir, Lamivudine, and the recommended phase 2 dose (RP2D) of Ritonavir determined in Part 1. Participants will receive up to 12 months of ART.
  Beginning Day 14 through Day 180, participants will receive adjuvant therapy, standard of care consisting of focal radiotherapy and Temozolomide therapy. Participants will receive focal radiotherapy for six weeks (42 days), and Temozolomide therapy, during and following radiotherapy up to Day 180.
  Participants will receive up to 12 months of study therapy, followed by up to 12 months of follow-up. Total participation duration is up to 24 months.
  Total participation is approximately two years.
  Interventions: Procedure: Magnetic Resonance (MR)-guided Laser Interstitial Thermal Therapy (LITT); Drug: Abacavir; Drug: Lamivudine; Drug: Ritonavir; Drug: Temozolomide; Radiation: Focal Radiotherapy

INTERVENTIONS:
Procedure: Magnetic Resonance (MR)-guided Laser Interstitial Thermal Therapy (LITT) — Participants will be administered MR-guided Laser Interstitial Thermal Therapy (LITT) as a single procedure, following stereotactic needle biopsy.
  Other Names: MR-Guided LITT
Drug: Abacavir — Participants will take one 600mg tablet of Abacavir orally once daily, as part of combination antiretroviral therapy (ART).
Drug: Lamivudine — Participants will take one 300mg tablet of Lamivudine orally once daily, as part of combination antiretroviral therapy (ART)
Drug: Ritonavir — Participants will take one tablet of Ritonavir (RTV) orally twice daily, as part of combination antiretroviral therapy (ART), at one of the following dose levels:
  * Dose Level 1: 100mg
  * Dose Level 2 (starting dose): 300mg
  * Dose Level 3: 400mg
  * Dose Level 4: 600mg
  Other Names: Norvir; RTV
Drug: Temozolomide — Participants will take Temozolomide (TMZ) via capsule orally, during and after focal radiotherapy, as part of standard of care adjuvant therapy. During focal radiotherapy, Temozolomide will be administered at a dose of 75 mg/m2 once daily for six weeks (42 days) on a continuous dosing regimen, including weekends and holidays. After completion of focal radiotherapy, Temozolomide will be administered at 150 mg/m^2 on days 1 through 5 of Cycle 1, and at 200 mg/m^2 on days 1 through 5 of Cycles 2 through 6, for a total of six 28-day cycles of maintenance therapy.
  Other Names: TMZ
Radiation: Focal Radiotherapy — Participants will be administered focal radiotherapy for six weeks (42 days), as part of adjuvant therapy, at a total dose of 50-60 grays (Gy) in 1.8-2.0 Gy fractions, depending on prognosis and as determined by the treating radiation oncologist.

SUMMARY:
The purpose of this study is to determine whether newly diagnosed high-grade glioma(s) that cannot be removed surgically change as a result of the study treatment; and to identify and evaluate the potential side effects (good and bad) of the study treatment in patients with newly diagnosed high-grade glioma(s) that cannot be removed surgically.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with a histologically confirmed or suspected high-grade glioma (HGG) by MRI.

   a. For cases with suspected HGG, intraoperative frozen section diagnoses of HGG must be made by pathologists (Section 4.4.1).
3. Uni-focal or butterfly gliomas that can receive ≥70% of lesion volume ablated as determined by the treating surgeon.
4. Gliomas must be located or positioned where surgical resection is either not feasible or high-risk as deemed by a group of surgical neuro-oncologists.
5. Preoperative Karnofsky score ≥ 70 (APPENDIX A).
6. Patients must have demonstrable normal organ function as defined below within 14 days of surgery.

   1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
   2. Platelets ≥ 100,000 cells/mm3
   3. Hemoglobin ≥ 9.0 g/dL. Use of transfusion or other intervention to achieve this hemoglobin level is acceptable.
   4. Blood urea nitrogen (BUN) ≤ 35 mg/dL and creatinine ≤ 1.9 mg/dL and estimated glomerular filtration rate (eGFR) or creatinine clearance rate > 50 mL per minute.
   5. Electrocardiogram (ECG) without evidence of acute cardiac ischemia.
   6. Prothrombin time (PT)/International Normalized Ratio (INR) <1.4
   7. Liver function tests: Aspartate aminotransferase (AST) and alanine transaminase (ALT) at or below 2.5 times the upper limit of normal (ULN).
   8. Sodium level > 130 mg/L. Use of salt resection or hypertonic saline to achieve this sodium level is acceptable.
7. Patients must be able to understand and sign informed consent.

Exclusion Criteria:

1. Patients with human leukocyte antigen (HLA) HLA-B*5701 hypersensitivity (Section 10.1.6.7).
2. Patients with sensitivity to abacavir, lamivudine, or ritonavir (Section 7.3.1).
3. Patients with a previous history of HIV infection.
4. Patients with uncontrolled hepatitis B or C infection.
5. Patients who have received any surgical resection for this tumor.

   a. Patients who have received an open biopsy for this disease are still eligible for participation.
6. Patients who have received chemotherapy or radiation for this disease.
7. Patients who are taking dofetilide (Section 4.10.1).
8. Patients on a regimen of 1 or more prohibited medications as described in Section 4.10.1 that cannot be discontinued or switched to a more compatible medication. For more information on prohibited and precautionary use medications for patients on this study, please see Section 4.10.
9. Patients not eligible to obtain MRI with and without contrast.
10. Recurrent HGG.
11. Presence of current infection, such as sepsis, meningitis, bacteremia, or pneumonia.
12. Fever within 48 hours of surgery (Temperature> 38.0°C).
13. Severe co-morbidity that would confer excess risk of surgery, radiation, or chemotherapy, as determined by the treating physician.
14. Any co-morbidity or psychiatric ailment that in the Investigator's opinion will prevent administration or completion of protocol therapy.
15. Pregnant women.
16. Patients must be willing to use contraception as described in Section 4.11.
17. Patients receiving other investigational agents or concurrent enrollment in another therapeutic clinical trial.
18. Prisoners.
19. Adults unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity | Up to 28 days
  The number of participants experiencing dose-limiting toxicity (DLT) during the first 28 days of antiretroviral therapy (ART) will be reported. Toxicity will be assessed by the treating physician and assigned severity and attribution using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).
Number of Participants Experiencing Serious Adverse Events and Grade 3 or Higher Adverse Events | Up to 12 months
  The number of participants experiencing serious adverse events (SAEs) and Grade 3 or higher adverse events (AEs) will be reported. SAEs and AEs will be assessed by the treating physician and assigned severity and attribution using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as percentage of participants without disease progression at time of study discontinuation.
Overall Survival (OS) | Up to 24 months
  Overall Survival is defined as the percentage of participants who are still living at the time of study discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Shah, MD, Principal Investigator — University of Miami; Macarena De La Fuente, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daftari M, Ramsoomair CK, Aaronson D, Seetharam D, Andreae EA, Wright L, Han S, Chandar J, Lu V, Govindarajan V, Ivan ME, Komotar RJ, de la Fuente M, Shah AH. Synergistic Treatment with Antiretrovirals and Laser Interstitial Thermal ThErapy (STARLITE) for unresectable glioblastoma: A phase 1 study protocol. PLoS One. 2025 Aug 28;20(8):e0328204. doi: 10.1371/journal.pone.0328204. eCollection 2025. PMID 40875628